CLINICAL TRIAL: NCT06580418
Title: Evaluation of an Anti-TREM-1 Treatment on an ex Vivo Human Intestinal Model
Acronym: TIME
Status: Recruiting | Type: Observational
Sponsor: Inotrem (Industry)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Sponsor
Other Study IDs: TIME
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Inflammatory Bowel Diseases
Keywords: IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ulcerative colitis (UC): 20 patients with moderate to severe UC under endoscopic surveillance for their disease
  Interventions: Other: Additional biopsies and blood samples
- Crohn's Disease (CD): 20 patients with moderate to severe CD under endoscopic surveillance for their disease
  Interventions: Other: Additional biopsies and blood samples

INTERVENTIONS:
Other: Additional biopsies and blood samples — During the endoscopic procedure planned for IBD patients following standard clinical practice, the endoscopist will decide the number and location of additional biopsy samples (up to 8) collected for the study. Participation in this study also requires the removal of three additional blood samples.

SUMMARY:
TIME is an observational study performed on UC and CD patients under endoscopic surveillance for monitoring the clinical activity of their disease.

The main objective of the study is to confirm the therapeutic potential of TREM-1 in inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 60 years
* Signed informed consent
* Ulcerative colitis (UC) patients with active disease
* Crohn's disease (CD) patients with active disease

Exclusion Criteria:

* UC or CD patients in remission
* Patients between 18 and 60 years without informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population that will be recruited for this study will be composed of patients with UC or CD under endoscopic surveillance for monitoring the clinical activity of their disease.
  The recruited patients will firstly sign the informed consent before undergoing the same day the blood withdrawal and endoscopy according to standard of care practice in the dedicated department, under the direction of the Gastroenterology and Digestive Endoscopy operative unit of the San Raffaele Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Collection of IBD patient-derived intestinal mucosal explants for testing TREM-1 antagonist | 20 months
  Derivation of RNA and proteins from biopsy specimens upon in vitro exposure to the TREM-1 antagonist

SECONDARY OUTCOMES:
Concentration of pro-inflammatory cytokines in supernatants of treated explants to evaluate the effect of the TREM-1 antagonist compound | 26 months
  Measurement of pro-inflammatory cytokine concentrations (pg/ml)
Gene expression in treated explants and other samples to evaluate the effect of the TREM-1 antagonist compound | 26 months
  RNAseq analysis

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No